CLINICAL TRIAL: NCT05232682
Title: Probiotics, Immune Function, and the Brain in Alcohol Consumers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2109003092; P01AA019072 (NIH)
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alcohol; Use, Problem
Keywords: alcohol use; probiotics; heavy drinking; brain; immune function
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Single group, open label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic Arm (Experimental): Probiotic arm
  Interventions: Dietary Supplement: Seed DS-01 Daily Synbiotic

INTERVENTIONS:
Dietary Supplement: Seed DS-01 Daily Synbiotic — Daily administration of Seed DS-01 Daily Synbiotic (dietary supplement)

SUMMARY:
This pilot project is a brief, open-label clinical trial of probiotics as an intervention in heavy drinkers. Heavy drinkers who do not yet show significant signs of liver disease may stand to benefit from probiotics, but no clinical trials to date have addressed this population. This study will recruit heavy drinkers to complete an open-label within-subjects trial. The study will investigate effects of probiotics on specific biomarkers in healthy heavy drinkers who currently are not seeking to change their alcohol use (i.e., are non-treatment-seeking).

DETAILED DESCRIPTION:
This pilot project is a brief, open-label clinical trial of probiotics as an intervention to reduce systemic and neural inflammation in heavy drinkers. Heavy drinkers who do not yet show significant signs of liver disease also may stand to benefit from probiotics, but no clinical trials to date have addressed this population. This study will recruit 15 non-treatment-seeking heavy drinkers to complete an open-label within-subjects trial. Aim 1 is to demonstrate proof-of-concept for beneficial effects of probiotic use on inflammatory processes. Aim 2 is to examine effects of probiotic use on brain metabolites correlated with neuroinflammation using magnetic resonance spectroscopy. Aim 3 is to gather preliminary data on acceptability and feasibility of the probiotic intervention in non-treatment-seeking heavy drinkers.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old;
* Able to speak and read English well enough to complete study procedures;
* Meets NIAAA guidelines for heavy drinking in the past 30 days.

Exclusion Criteria:

* Chronic disease requiring daily use of medication;
* Seeking or receiving treatment for alcohol/drug use, with exception of smoking cessation;
* Self-reported history of liver disease;
* Antibiotic or probiotic use in past 1 month;
* Positive urine drug test;
* History of fainting, weakness, infection, excessive bruising, or extreme distress from blood draw;
* Safety contraindication for MRI (e.g., ferromagnetic implant in the body, claustrophobia);
* Head trauma with loss of consciousness >10 min;
* Pregnant, breastfeeding, or not using effective birth control;
* Unable to complete the study visits due to time or scheduling constraints;
* Weight <110 lbs.
* Conditions of immunodeficiency, such as HIV infection, primary immune deficiency, or taking immune-suppressant medications.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mollie Monnig, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants from February 2022 to November 2022. Participants were recruited from the Providence, Rhode Island, area using flyers and online advertising.
Pre-assignment Details: Of 32 participants enrolled for initial screening, 16 participants were fully eligible for the study after Visit 1 assessment and initiated the probiotic course. Two participants were lost to follow-up prior to completing the probiotic course. Fourteen participants completed the 30-day follow-up visit.
Period: Overall Study
Arm/Group | Probiotic Arm
Started | 16
Completed | 14
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Probiotic Arm
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Participants were recruited from the greater Providence area in Rhode Island, USA.
  participants
    United States | 16
Number of drinks in past 30 days [Mean (Standard Deviation); unit: US standard drinks] | 66.2 (33.5)

OUTCOME MEASURES:

1. Primary Outcome: Lipopolysaccharide Binding Protein (LBP)
Description: LBP levels in plasma
Time Frame: 30 days: Probiotic Arm is baseline; Probiotic Arm at Follow-up is the 30-day follow-up data on the same group.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Probiotic Arm: Probiotic arm at baseline
  Seed DS-01 Daily Synbiotic: Daily administration of Seed DS-01 Daily Synbiotic (dietary supplement)
- Probiotic Arm at Follow-Up: Probiotic Arm within subjects at 30-day follow-up
Arm/Group | Probiotic Arm | Probiotic Arm at Follow-Up
Number analyzed (Participants) | 16 | 14
ng/ml | 23609.2 (11451.8) | 28111.9 (16621.6)
Statistical Analysis 1: Comparison: Probiotic Arm vs Probiotic Arm at Follow-Up; Test type: Other; p = 0.1183, Mixed Models Analysis — Alpha value for significance set at p < .05; F-test = 2.41

2. Primary Outcome: Soluble Cluster of Differentiation 14 (sCD14)
Description: sCD14 levels in plasma
Time Frame: 30 days: Probiotic Arm is baseline; Probiotic Arm at Follow-up is the 30-day follow-up data on the same group.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Probiotic Arm | Probiotic Arm at Follow-Up
Number analyzed (Participants) | 16 | 14
ng/ml | 3175.9 (1577.3) | 3394.7 (1973.2)
Statistical Analysis 1: Comparison: Probiotic Arm vs Probiotic Arm at Follow-Up; Test type: Other; p = 0.9308, Mixed Models Analysis — Alpha value for significance set at p < .05; F-test = 0.07

3. Primary Outcome: Soluble Cluster of Differentiation 163 (sCD163)
Description: sCD163 levels in plasma
Time Frame: 30 days: Probiotic Arm is baseline; Probiotic Arm at Follow-up is the 30-day follow-up data on the same group.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Probiotic Arm | Probiotic Arm at Follow-Up
Number analyzed (Participants) | 16 | 14
ng/ml | 518.6 (288.1) | 560.9 (205.2)
Statistical Analysis 1: Comparison: Probiotic Arm vs Probiotic Arm at Follow-Up; Test type: Other; p = 0.1517, Mixed Models Analysis — Alpha value for significance set at p < .05; F-test = 2.10

4. Primary Outcome: Interleukin-6 (IL-6)
Description: IL-6 levels in plasma
Time Frame: 30 days: Probiotic Arm is baseline; Probiotic Arm at Follow-up is the 30-day follow-up data on the same group.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Probiotic Arm | Probiotic Arm at Follow-Up
Number analyzed (Participants) | 16 | 14
pg/ml | 1.2 (0.8) | 1.2 (0.6)
Statistical Analysis 1: Comparison: Probiotic Arm vs Probiotic Arm at Follow-Up; Test type: Other; p = 0.8747, Mixed Models Analysis — Alpha value for significance set at p < .05; F-test = 0.14

5. Primary Outcome: Monocyte Chemoattractant Protein-1 (MCP-1)
Description: MCP-1 levels in plasma
Time Frame: 30 days: Probiotic Arm is baseline; Probiotic Arm at Follow-up is the 30-day follow-up data on the same group.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Probiotic Arm | Probiotic Arm at Follow-Up
Number analyzed (Participants) | 16 | 14
pg/ml | 93.5 (24.4) | 101.0 (22.8)
Statistical Analysis 1: Comparison: Probiotic Arm vs Probiotic Arm at Follow-Up; Test type: Other; p = 0.3269, Mixed Models Analysis — Alpha value for significance set at p < .05; F-test = 1.19

6. Primary Outcome: Tumor Necrosis Factor Alpha (TNF-a)
Description: TNF-a levels in plasma
Time Frame: 30 days: Probiotic Arm is baseline; Probiotic Arm at Follow-up is the 30-day follow-up data on the same group.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Probiotic Arm | Probiotic Arm at Follow-Up
Number analyzed (Participants) | 16 | 14
pg/ml | 7.4 (0.9) | 7.6 (1.8)
Statistical Analysis 1: Comparison: Probiotic Arm vs Probiotic Arm at Follow-Up; Test type: Other; p = 0.3411, Mixed Models Analysis — Alpha value for significance set at p < .05; F-test = 1.14

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Probiotic Arm
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT05232682/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT05232682/ICF_001.pdf